CLINICAL TRIAL: NCT01522170
Title: An Observational, Multi-Center, Multi-National, Long Term Follow-Up Study of Atypical Hemolytic Uremic Syndrome (aHUS) Patients Treated With Eculizumab in a Prior Clinical Study
Brief Title: aHUS Observational Long Term Follow-Up
Acronym: LTFU
Status: Terminated | Type: Observational
Why Stopped: Remaining patients were offered a similar observational study (Alexion M11-001) to allow for robust, high quality data collection in a larger, single database
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C11-003
Record Dates: First submitted 2012-01-18; First posted 2012-01-31 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Atypical Hemolytic Uremic Syndrome
Keywords: Atypical Hemolytic Uremic Syndrome; aHUS; Eculizumab
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
There is growing but limited information on the long term clinical status of aHUS patients who have previously received or are continuing to receive treatment with eculizumab. This study is designed to collect clinical data that will provide insight into the long-term outcomes of patients with aHUS.

ELIGIBILITY:
Inclusion Criteria:

* aHUS patients who participated in any one of the aHUS-eculizumab clinical studies.
* aHUS patients or legal representative who are able and willing to given written informed consent for their study information to be collected and retained in a database.

Exclusion Criteria:

* Not applicable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female aHUS, including minors, who previously participated in eculizumab clinical trials.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
TMA complication-free survival | 5 Years
  Assess the long term efficacy of eculizumab in patients with aHUS who have previously participated in an eculizumab clinical study.

SECONDARY OUTCOMES:
Duration of response, change over time of value for platelets, LDH, eGFR, Hgb, TMA intervention | 5 Years
  Assess the long term safety of eculizumab in patients with aHUS who have previously participated in an eculizumab clinical study by collecting data on serious adverse events and targeted adverse events.

CONTACTS AND LOCATIONS:
Locations (56):
- United States (16):
  - Emory Healthcare - Children's Center, Atlanta, Georgia
  - Dunwoody Pediatrics & Children's Healthcare of Atlanta, Dunwoody, Georgia
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Fort Wayne, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Hudson Valley Oncology Hematology, Hawthorne, New York
  - Weill Cornell Medical College, New York, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Arthur James Cancer Hospital, Columbus, Ohio
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center & Children's Hospital, Spokane, Washington
  - Fox Valley Hematology, Oshkosh, Wisconsin
- Royal Adelaide Hospital, North Tce. Adelaide, Australia
- Austria (2):
  - Universitatsklinik fur Innere Medizin Medizinische Universitat Graz, Graz
  - Medizinische Universitaet Innsbruck, Innsbruck
- Belgium (2):
  - UZ Gent Dienst nefrologie, Ghent
  - Chu Sart Tilman, Liège
- Canada (2):
  - Centre Hospitalier Universitaire (CHU) Sainte-Justine, Montreal
  - The Hospital for Sick Children, Toronto
- France (17):
  - Centre Hospitalier Universitaire Pellegrin, Service de Nephrologie Transplantation Dialyse, Bordeaux
  - CHRU de Caen, Caen
  - Le Kremlin Bicetre Hospital, Nephrology Unit, Le Kremlin-Bicêtre
  - CHRU de Lille-Hopital A.Calmette, Lille
  - Hôpital Edouard Herriot, Lyon
  - Hopital de la Timone Enfants, Unité de Néphrologie, Marseille
  - CHU Hotel Dieu, Nantes
  - Le Centre Hospitalier Universitaire de Nice, Nice
  - Centre Hospitalier Regional de la Source, Service de nephrologie/hemodialyse, Orléans
  - Hopital Robert-Debré, Service de Néphrologie Pédiatrique, Paris
  - Hopital Tenon, Paris
  - Centre Hospitalier Inter-Communal de Cornouaille, Quimper
  - CHU-CH Charles Nicolle Pavillon de Pédiatrie, Rouen
  - Hôpital de Bois Guillaume CHU de Rouen, Rouen
  - CHU de Saint-Etienne, Saint-Priest-en-Jarez
  - Nouvel Hopital Civil, Strasbourg
  - CHRU de Tours, Tours
- Germany (3):
  - Universitaetsklinikum Aachen Klinik fuer Nieren- und Hochdruckkrankheiten, Aachen
  - Hannover University Clinic, Hanover
  - Universitaet Heidelberg, Heidelberg
- Italy (5):
  - A.O. Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Istituto Giannina Gaslini, Genova
  - Fondazione IRCCS Ca Granda, Ospedale Maggiore Policlinico Maggiore Policlinico, Milan
  - Ospedale dei Bambini G. di Cristina, Palermo
- Netherlands (2):
  - AMC Medical Research B.V., Amsterdam
  - Radboud University Nijmegen Medical Centre Nijmegen, Nijmegen
- Nephrology Clinic, Karolinska University Hospital, Stockholm, Sweden
- INSELSPITAL Universitaetsklinik fuer Kinderheilkunde Kindernephrologie, Bern, Switzerland
- United Kingdom (4):
  - Royal Devon & Exeter NHS Foundation Trust, Exeter
  - Gartnavel General Hospital, Glasgow
  - The Newcastle upon Tyne Hospitals NHS, Newcastle upon Tyne
  - City Hospital, Nottingham University Hospitals, NHS Trust, Nottingham

REFERENCES:
- [Derived] Menne J, Delmas Y, Fakhouri F, Licht C, Lommele A, Minetti EE, Provot F, Rondeau E, Sheerin NS, Wang J, Weekers LE, Greenbaum LA. Outcomes in patients with atypical hemolytic uremic syndrome treated with eculizumab in a long-term observational study. BMC Nephrol. 2019 Apr 10;20(1):125. doi: 10.1186/s12882-019-1314-1. PMID 30971227